CLINICAL TRIAL: NCT07286474
Title: The Effects of Combined Low-Level Laser Therapy (LLLT) and Oral Vitamin D3 Supplements on Orthodontic Tooth Movements: A Randomized Controlled Trial.
Brief Title: Effects of Laser Therapy and Vitamin D Pills on Braces Tooth Movement: A Random Controlled Study
Acronym: LLLT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Syed Abid Altaf Bukhari, PhD Student, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/24040356
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Malocclusion of Anterior Teeth
Keywords: LLLT, vitamin D3 supplements, randomized controlled trial, mandibular crowding, root resorption, pain perception, acceleration of orthodontics
MeSH Terms: conditions — Root Resorption | interventions — Cholecalciferol; Low-Level Light Therapy; Orthodontic Appliances, Fixed

STUDY DESIGN:
Intervention Model Description: The three study arms in this randomized controlled trial are as follows:
  * Group 1A (Experimental): Standard orthodontic treatment (braces) plus oral Vitamin D3 supplements (initial 50,000 IU dose one week before treatment, followed by 1,000 IU daily maintenance).
  * Group 1B (Experimental): Standard orthodontic treatment (braces) plus oral Vitamin D3 supplements (as above) combined with Low-Level Laser Therapy (LLLT) applied to the gums at specified intervals.
  * Control Group: Standard orthodontic treatment (braces) only, with no Vitamin D3 supplements or LLLT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vitamin D3 Only Group (Experimental): Participants receive standard orthodontic treatment with pre-adjusted edgewise brackets (0.022" MBT prescription) and wire sequencing (0.014" NiTi initial, progressing to 0.017x0.025" SS). Additionally, oral Vitamin D3 supplementation: single loading dose of 50,000 IU one week before treatment, followed by 1,000 IU daily maintenance until alignment completion. No LLLT.
  Interventions: Dietary Supplement: Cholecalciferol (Vit D3); Device: Fixed Orthodontic Appliance
- Vitamin D3 + LLLT Group (Experimental): Participants receive standard orthodontic treatment as above. Plus oral Vitamin D3 supplementation (50,000 IU loading one week before, 1,000 IU daily). Plus LLLT using InGaAlAs diode laser (940 nm, 2.5 W, 25.7 J/cm², 30 seconds labially at muco-gingival junction) initiated at alignment start, repeated on days 14 and 30, then every 4 weeks until completion.
  Interventions: Dietary Supplement: Cholecalciferol (Vit D3); Radiation: Low-Level Laser Therapy
- Control Group (Active Comparator): Participants receive only standard orthodontic treatment with pre-adjusted edgewise brackets (0.022" MBT prescription) and wire sequencing (0.014" NiTi initial, progressing to 0.017x0.025" SS). No Vitamin D3 supplementation or LLLT.
  Interventions: Device: Fixed Orthodontic Appliance

INTERVENTIONS:
Dietary Supplement: Cholecalciferol (Vit D3) — Oral cholecalciferol supplementation: initial loading dose of 50,000 IU one week before orthodontic treatment initiation, followed by daily maintenance dose of 1,000 IU until alignment completion. Administered to participants with baseline sufficient Vitamin D levels.
  Arms: Vitamin D3 + LLLT Group; Vitamin D3 Only Group
Radiation: Low-Level Laser Therapy — Diode laser (Biolase 10W 940±10nm, InGaAlAs) with tooth whitening handpiece (spot size 2.8 cm²), wavelength 940 nm, power output 2.5 W, energy density 25.7 J/cm², continuous wave mode. Applied labially in direct contact at mucogingival junction for 30 seconds. Initiated at alignment start, repeated on days 14 and 30, then every 4 weeks until completion. Eye protection worn by operator and participant.
  Arms: Vitamin D3 + LLLT Group
Device: Fixed Orthodontic Appliance — Pre-adjusted edgewise conventional brackets with 0.022" MBT (McLaughlin Bennett Trevisi) prescription (3M Unitek), bondable 0.022" single slot molar tubes, bonded using Transbond XT light cure material on upper and lower arches. Wire sequencing: initial 0.014" super elastic nickel-titanium (SE-NiTi), followed by 0.016" SE-NiTi, 0.016 x 0.022" SE-NiTi, and finally 0.017 x 0.025" stainless steel wire until alignment completion. Adjustments every 4 weeks.
  Arms: Control Group; Vitamin D3 Only Group

SUMMARY:
This clinical trial aims to evaluate the efficacy of low-level laser therapy (LLLT) in conjunction with oral vitamin D3 supplementation in accelerating orthodontic tooth movement in adults with crowded mandibular anterior teeth undergoing orthodontic treatment. Additionally, the study seeks to assess the safety profile and potential adverse effects, including pain and root resorption.

The primary research questions are as follows:

1. Does vitamin D3 enhance the rate of orthodontic tooth movement?
2. Does the combination of vitamin D3 and LLLT result in a greater acceleration of tooth movement compared to either intervention alone?
3. Do vitamin D3 and LLLT influence the extent of root resorption?
4. Do vitamin D3 and LLLT mitigate pain associated with orthodontic treatment?
5. Do vitamin D3 and LLLT reduce the frequency of required clinical visits?

The study will compare the outcomes of orthodontic treatment with braces alone, braces with vitamin D3 supplementation, and braces with both vitamin D3 and LLLT, to determine their effects on the rate of tooth movement, pain reduction, and root resorption.

Participants will undergo the following procedures:

* A blood test to assess baseline vitamin D levels.
* Placement of orthodontic braces.
* Daily administration of vitamin D3 supplements for those assigned to the relevant groups, commencing with a loading dose one week prior to the initiation of orthodontic treatment.
* Application of LLLT to the gingival tissues for participants in the corresponding group, administered at the start and during follow-up visits.
* Regular clinic visits every four weeks for monitoring, pain assessment, and measurement of tooth movement until the completion of orthodontic alignment.

DETAILED DESCRIPTION:
Orthodontic treatment is instrumental in aligning teeth and enhancing both aesthetic and functional aspects of smiles and bites. However, the duration of such treatment is typically protracted, averaging between 1.5 to 3 years. This extended timeframe can result in complications such as discomfort, root resorption, plaque accumulation, periodontal issues, and enamel demineralization. Both patients undergoing orthodontic treatment and their orthodontists seek methods to expedite the process without compromising safety. Orthodontic tooth movement is facilitated by the application of gentle forces through Standard Orthodontic treatment , which induce remodeling of the surrounding bone. This process involves bone resorption on one side and new bone formation on the other, mediated by osteoclasts and osteoblasts, as well as the involvement of blood vessels and nerves within the periodontal tissues. Over time, various strategies have been explored to accelerate tooth movement. Surgical interventions, such as corticotomy or piezocision, have demonstrated efficacy in hastening the process but are invasive and may cause apprehension among patients. Non-surgical approaches, including vibrational devices, magnetic fields, or hormonal injections, have been investigated, though some present adverse effects or limited efficacy. Low-level laser therapy (LLLT) emerges as a non-invasive alternative, utilizing low-energy light to enhance healing processes. LLLT has been shown to augment blood circulation, reduce inflammation, and enhance the function of bone cells. Empirical evidence suggests that LLLT may accelerate orthodontic tooth movement by modulating proteins and cellular activities involved in bone remodeling, such as increasing RANKL expression, which facilitates bone resorption, and alleviating orthodontic pain.

Vitamin D3, commonly referred to as the "sunshine vitamin," is essential for maintaining bone health. It is synthesized in the body through skin exposure to sunlight or obtained from dietary sources such as fish, eggs, or supplements. Vitamin D3 plays a crucial role in regulating calcium and phosphorus levels, which are vital for strong bones. In the field of orthodontics, vitamin D3 may facilitate bone remodeling during tooth movement. Animal studies have indicated that local injections of vitamin D3 near teeth can enhance movement; however, human studies have yielded mixed results, with some demonstrating accelerated movement with local vitamin D3 application, while others do not. Oral supplementation is considered safer and more convenient, yet there is a paucity of research examining its effects on orthodontic treatment. To date, no studies have investigated the combined use of low-level laser therapy (LLLT) and oral vitamin D3. It is hypothesized that these interventions may have a synergistic effect: vitamin D3 enhances bone metabolism, while LLLT reduces inflammation and promotes healing. This study aims to address this gap by evaluating whether the combination of LLLT and oral vitamin D3 accelerates the alignment of crowded lower anterior teeth more effectively than either treatment alone, while also monitoring potential side effects such as pain or root resorption.

This study is a randomized controlled trial comprising three groups to facilitate an equitable comparison of treatments. The participants are adults aged 18 to 40 years, exhibiting moderate dental crowding (4-8 mm) in the mandibular anterior region, necessitating orthodontic intervention. Eligibility criteria include normal vitamin D levels, overall good health, and a complete set of permanent teeth. Exclusion criteria encompass individuals with deficient vitamin D levels, specific medical conditions (such as thyroid or renal disorders), pregnancy, or inadequate oral hygiene. The target sample size is approximately 39 participants, distributed equally among the groups: Group A will receive orthodontic Standard Orthodontic treatment in conjunction with daily vitamin D3 supplementation, beginning with a high dose followed by maintenance dosing; Group B will receive Standard Orthodontic treatment , vitamin D3 supplementation, and low-level laser therapy (LLLT); the Control Group will receive Standard Orthodontic treatment only. Randomization is conducted using software to mitigate bias. The study adheres to ethical standards and the CONSORT guidelines to ensure transparent reporting.Procedures Initially, all participants undergo blood tests to assess vitamin D levels. Individuals with deficient levels are referred for treatment and are excluded from participation. Eligible participants provide informed consent and undergo standard orthodontic documentation, including photographs, X-rays, and study models. The orthodontic treatment commences with the application of 0.022" MBT-type Standard Orthodontic treatment on both the upper and lower dentition. The orthodontic wires are incrementally thickened to facilitate dental alignment, beginning with 0.014" flexible nickel-titanium, followed by 0.016", 0.016x0.022", and ultimately 0.017x0.025" steel wires. For the vitamin D3 cohort, a 50,000 IU dose is administered one week prior to the initiation of orthodontic treatment, followed by a daily intake of 1,000 IU until dental alignment is achieved. In the Low-Level Laser Therapy (LLLT) group, a diode laser (940 nm, 2.5 W power) equipped with a whitening handpiece is employed. The laser light is applied directly to the gingival tissue above the lower anterior teeth for 30 seconds at the commencement of treatment, on day 14, day 30, and subsequently every four weeks. Protective eyewear is mandatory during these sessions. Progress evaluations occur at four-week intervals, utilizing Little's Irregularity Index on study models to quantify dental crowding by summing the interproximal contact point discrepancies of the lower anterior teeth. Treatment concludes when the index reaches 0 mm, indicating complete alignment. Root resorption is assessed through comparative pre- and post-treatment X-rays of the lower anterior teeth, graded on a scale from 0 (no change) to 4 (severe resorption). Pain levels are documented daily for seven days following each wire adjustment or laser session, using a 10-cm visual analog scale (0 indicating no pain, 10 indicating the most severe pain). Participants also record any analgesic consumption. Data analysis involves statistical tests to compare the groups regarding treatment duration, root resorption, and pain levels. The findings have the potential to inform the development of more efficient and less painful orthodontic treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

Participants requiring orthodontic treatment for crowding in the range of 4 to 8 mm in the lower anterior segment.

• Age range: 18 to 40 years.

• Angles Class I, II or III malocclusion

• Fully erupted permanent dentition

• Good oral and general health

- Normal range of Vitamin D levels

Exclusion Criteria:

* Deficiency of Vitamin D levels below normal range. • Medically compromised patients with thyroid, parathyroid, or renal and liver diseases.

Patients on medication, especially corticosteroid and anticonvulsant drugs • Poor oral hygiene

• Pregnancy

• Lactation

• History of craniofacial abnormalities or syndromes that may affect orthodontic tooth movements.

• Participants failing to complete the Vitamin D supplementation log sheets will be excluded to ensure accurate data collection.

• Inability to comply with the study protocol or unable to complete the study due to personal, medical, or logistical reasons (e.g., missed follow-up visits or failure to undergo assessments) will be excluded to maintain data integrity and minimize biases from incomplete participation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Orthodontic Tooth Movement | From baseline (initiation of alignment) to complete alignment (Little's Irregularity Index reaches 0 mm), assessed every 4 weeks (estimated duration 6-10 months per participant)
  The rate of reduction in mandibular anterior crowding, measured in mm/month using Little's Irregularity Index (sum of linear displacements between contact points of the six mandibular anterior teeth from canine to canine, assessed via dental models). Compared across groups to evaluate acceleration effects.

SECONDARY OUTCOMES:
Root Resorption | Baseline and at completion of alignment (estimated 6-10 months)
  Degree of apical root resorption in mandibular anterior teeth, assessed using periapical radiographs and graded on a 0-4 scale (0 = no resorption, 4 = severe resorption >4 mm). Compared between baseline and post-alignment images.
Pain Perception | Daily for 7 days after each monthly visit, throughout the alignment phase (up to 10 months)
  Orthodontic pain intensity measured using a 10-cm Visual Analogue Scale (VAS; 0 = no pain, 10 = worst pain imaginable). Participants record daily scores for 7 days following each archwire activation or LLLT session.
Duration of Orthodontic Alignment | From baseline to complete alignment, monitored every 4 weeks (estimated 6-10 months)
  Total time required to achieve complete resolution of mandibular anterior crowding (from initiation of fixed appliance treatment to Little's Irregularity Index of 0 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Rozita Hassan, BDS, MS, MOrtho RCSEd, Study Director — Universiti Sains Malayisa
Locations (1):
- Armed Forces Hospital, Madinah, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No